CLINICAL TRIAL: NCT04856007
Title: A Single-centre, Parallel-cohort, Randomized, Open-label, Two-period, Cross-over, Bioequivalence Study of the Fixed Dose Combination of Dapagliflozin/Metformin XR Relative to Co-administration of the Individual Components in Two Cohorts of Healthy Chinese Subjects in the Fed State.
Brief Title: A Study to Assess the Bioequivalence of Fixed Dose Combination of Dapagliflozin/Metformin XR Relative to Co-administration of the Individual Components in Healthy Chinese Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: D1691C00011
Record Dates: First submitted 2021-04-09; First posted 2021-04-22 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteer
Keywords: Dapagliflozin; Forxiga; Metformin XR; Glucophage XR; Xigduo XR; Bioequivalence; Cross-over
MeSH Terms: interventions — dapagliflozin; Metformin

STUDY DESIGN:
Intervention Model Description: There will be two independent cohorts of subjects who will each receive two treatments in a randomized order, and each treatment will be followed by 72 hours of blood sampling for pharmacokinetic assessments, with safety and tolerability. In each cohort approximately 40 healthy subjects will be randomized to receive treatment with IP in order to complete at least 36 evaluable subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dapagliflozin 5mg + Metformin 500mg XR (Experimental): co-administration of a single oral dose of a 5mg dapagliflozin (Forxiga® 5mg) tablet and a 500mg metformin XR (Glucophage XR®) tablet
  Interventions: Drug: Dapagliflozin/metformin XR FDC 5/500 mg
- Dapagliflozin/metformin XR FDC 5/500 mg (Experimental): single FDC tablet consisting of 5mg dapagliflozin and 500mg metformin XR subject
  Interventions: Drug: Dapagliflozin 5 mg + Metformin 500 mg XR
- Dapagliflozin 10mg + Metformin 1000mg XR (Experimental): co-administration of a single oral dose of a 10mg dapagliflozin (Forxiga® 10mg) tablet and two 500mg metformin XR (Glucophage XR®) tablets
  Interventions: Drug: Dapagliflozin/metformin XR FDC 10/1000 mg
- Dapagliflozin/metformin XR FDC 10/1000 mg (Experimental): ingle FDC tablet consisting of 10mg dapagliflozin and 1000mg metformin XR
  Interventions: Drug: Dapagliflozin 10 mg + Metformin 1000 mg XR

INTERVENTIONS:
Drug: Dapagliflozin/metformin XR FDC 5/500 mg — In cohort 1, subjects will be randomized to receive co-administration of a single oral dose of a 5mg dapagliflozin tablet and a 500mg metformin XR tablets (Treatment A) followed by 7 to 14 days washout and then receive single FDC tablet consisting of 5mg dapagliflozin and 500mg metformin XR (Treatment B) on Day 1 in one treatment sequence. Or subjects will be randomized to be administered the Treatment B followed by 7 to 14 days washout and then received Treatment A on Day1 in the other treatment sequence.
  Other Names: Xigduo XR
  Arms: Dapagliflozin 5mg + Metformin 500mg XR
Drug: Dapagliflozin/metformin XR FDC 10/1000 mg — In cohort 2, subjects will be randomized to receive co-administration of a single oral dose of a 10mg dapagliflozin tablet and two 500mg metformin XR tablets (Treatment C) followed by 7 to 14 days washout and then receive single FDC tablet consisting of 10mg dapagliflozin and 1000mg metformin XR (Treatment D) on Day 1 in one treatment sequence. Or subjects will be randomized to be administered the Treatment D followed by 7 to 14 days washout and then received Treatment C on Day1 in the other treatment sequence.
  Other Names: Xigduo XR
  Arms: Dapagliflozin 10mg + Metformin 1000mg XR
Drug: Dapagliflozin 5 mg + Metformin 500 mg XR — In cohort 1, subjects will be randomized to receive co-administration of a single oral dose of a 5mg dapagliflozin tablet and a 500mg metformin XR tablets (Treatment A) followed by 7 to 14 days washout and then receive single FDC tablet consisting of 5mg dapagliflozin and 500mg metformin XR (Treatment B) on Day 1 in one treatment sequence. Or subjects will be randomized to be administered the Treatment B followed by 7 to 14 days washout and then received Treatment A on Day1 in the other treatment sequence.
  Other Names: Forxiga + Glucophage XR
  Arms: Dapagliflozin/metformin XR FDC 5/500 mg
Drug: Dapagliflozin 10 mg + Metformin 1000 mg XR — In cohort 2, subjects will be randomized to receive co-administration of a single oral dose of a 10mg dapagliflozin tablet and two 500mg metformin XR tablets (Treatment C) followed by 7 to 14 days washout and then receive single FDC tablet consisting of 10mg dapagliflozin and 1000mg metformin XR (Treatment D) on Day 1 in one treatment sequence. Or subjects will be randomized to be administered the Treatment D followed by 7 to 14 days washout and then received Treatment C on Day1 in the other treatment sequence.
  Other Names: Forxiga + Glucophage XR
  Arms: Dapagliflozin/metformin XR FDC 10/1000 mg

SUMMARY:
To assess the bioequivalence between dapagliflozin/metformin XR FDC tablet and co-administration of dapagliflozin and metformin XR tablets.

DETAILED DESCRIPTION:
A Single-centre, Parallel-cohort, Randomized, Open-label, Two-period, Cross-over, Bioequivalence Study of the Fixed Dose Combination of Dapagliflozin/Metformin XR Relative to Co-administration of the Individual Components in Two Cohorts of Healthy Chinese Subjects in the Fed State.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures.
2. Healthy Chinese subjects as determined by no clinically significant deviation from normal in medical history, vital signs, physical examination, 12-lead ECG, and clinical laboratory evaluations.
3. Male or female, ages 18 to 55 years, inclusive, at the time of signing the informed consent
4. Weigh at least 50 kg (for male) and 45 kg (for female), respectively, and have a body mass index (BMI) ≥ 19 and <26 kg/m2. BMI = weight (kg)/[height (m)]2.
5. Female participants: Women of childbearing potential must use one highly effective form of birth control.
6. Must be able to communicate with the investigator, understand and comply with all study requirements.

Exclusion Criteria:

1. Any significant acute or chronic medical illness.
2. Current or recent (within 3 months prior to study drug administration) gastrointestinal disease that may impact drug absorption and affect PK of the study drugs. Additionally, any gastrointestinal surgery (eg, partial gastrectomy, pyloroplasty) that could impact the absorption of study drug.
3. Any major surgery, as determined by the investigator, within 4 weeks prior to study drug administration.
4. Donation of blood within 3 months prior to study drug administration.
5. Blood transfusion within 4 weeks prior to study drug administration.
6. Inability to tolerate oral medication.
7. Inability to tolerate venous access.
8. Drug or alcohol abuse within 6 months prior to study drug administration. Alcohol abuse is defined as a history of regular alcohol consumption exceeding 14 drinks per week, or a positive breath alcohol test at screening and/or check-in. 1 drink equals to 5 ounces (150ml) of wine or 12 ounces (360 ml) of beer or 1.5 ounces (45 ml) of hard liquor.
9. Regularly drink more than 3 cups of coffee or other caffeine-containing products a day, or 5 cups of tea a day.
10. Regular smoker (the subject should be able to abstain from smoking for the duration of the study without having abstinence, therefore they should not be regular smokers, regular smokers are defined as people who smoke everyday), use of tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 4 weeks prior to study drug administration .
11. Any other sound medical, psychiatric and/or social reason as determined by the investigator.
12. Any of the following on ECG prior to study drug administration:

    1. PR≥210ms
    2. QRS≥120ms
    3. QT≥500ms
    4. QTcF≥450ms(male) or QTcF≥470ms(female)
13. Positive urine screen for drugs of abuse.
14. Any clinically significant abnormal findings in urinalysis (may repeat once) at screening, as judged by the investigator.
15. Glucosuria at screening.
16. Abnormal liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], or total bilirubin > 10% above upper limit of normal [ULN]).
17. Elevated serum creatinine (> ULN).
18. Positive blood screen for HIV antibody , Syphilis antibody, hepatitis C antibody , or Hepatitis B surface antigen (HbsAg) or only Hepatitis B core antibody (anti-HBc) in Hepatitis B serologic test.
19. History of allergy to SGLT2 inhibitor drug class or related compounds.
20. History of allergy or intolerance to metformin or other similar acting agents.
21. History of any significant drug allergy (such as anaphylaxis or hepatotoxicity).
22. Prior exposure to metformin or dapagliflozin within 3 months of study drug administration.
23. Exposure to any investigational product or placebo within 4 weeks prior to study drug administration.
24. Use of any prescription drugs or over-the counter (OTC), traditional Chinese medicine and herbal preparations within 4 weeks prior to study drug administration.
25. Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff or staff at the study site).
26. Previous enrolled or randomized in the present study.
27. For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.
28. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
29. Has clinical signs and symptoms consistent with COVID-19 infection (eg fever, dry cough, dyspnea, sore throat, fatigue.. etc) as judged by investigator or confirmed infection by appropriate laboratory test within the last 4 weeks prior to screening or on admission.
30. History of COVID-19.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from zero to the last quantifiable concentration(AUClast) of dapagliflozin and metformin. | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  For period 1 and 2, PK samples will be collected pre-dose and 0.5,1,2,3,4,6,8,10,12,24(Day2),36,48(Day3), and 72(Day4) hours post dose.
Area under the plasma concentration-time curve from zero to infinity (AUCinf) of dapagliflozin and metformin. | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  For period 1 and 2, PK samples will be collected pre-dose and 0.5,1,2,3,4,6,8,10,12,24(Day2),36,48(Day3), and 72(Day4) hours post dose.
Maximum observed plasma concentration (Cmax) of dapagliflozin and metformin. | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  For period 1 and 2, PK samples will be collected pre-dose and 0.5,1,2,3,4,6,8,10,12,24(Day2),36,48(Day3), and 72(Day4) hours post dose.

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration (tmax) of dapagliflozin and metformin. | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  For period 1 and 2, PK samples will be collected pre-dose and 0.5,1,2,3,4,6,8,10,12,24(Day2),36,48(Day3), and 72(Day4) hours post dose.
Terminal elimination rate constant (λz) of dapagliflozin and metformin. | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  For period 1 and 2, PK samples will be collected pre-dose and 0.5,1,2,3,4,6,8,10,12,24(Day2),36,48(Day3), and 72(Day4) hours post dose.
Half-life associated with terminal slope of a semi-logarithmic concentration-time curve(t½λz) of dapagliflozin and metformin. | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  For period 1 and 2, PK samples will be collected pre-dose and 0.5,1,2,3,4,6,8,10,12,24(Day2),36,48(Day3), and 72(Day4) hours post dose.
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) of dapagliflozin and metformin. | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  For period 1 and 2, PK samples will be collected pre-dose and 0.5,1,2,3,4,6,8,10,12,24(Day2),36,48(Day3), and 72(Day4) hours post dose.
Apparent volume of distribution following extravascular administration (Vz/F) of dapagliflozin and metformin. | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  For period 1 and 2, PK samples will be collected pre-dose and 0.5,1,2,3,4,6,8,10,12,24(Day2),36,48(Day3), and 72(Day4) hours post dose.

OTHER OUTCOMES:
Haematology and clinical chemistry laboratory variables over time - SI unit - Change from baseline | Day 2 and Day 4 in Treatment period 1 and 2, respectively.
  To further assess the safety and tolerability of dapagliflozin/metformin XR FDC and coadministration of the individual components in healthy Chinese subjects in the fed state.
Vital signs over time - Change from baseline | From Day 2 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  To further assess the safety and tolerability of dapagliflozin/metformin XR FDC and coadministration of the individual components in healthy Chinese subjects in the fed state.
ECG variables over time - Change from baseline | Day 1, 4 hours and 8 hours after dosing and Day 4 in Treatment period 1 and 2, respectively.
  To further assess the safety and tolerability of dapagliflozin/metformin XR FDC and coadministration of the individual components in healthy Chinese subjects in the fed state.
Urinalysis data over time | Day 2 and Day 4 in Treatment period 1 and 2, respectively.
  To further assess the safety and tolerability of dapagliflozin/metformin XR FDC and coadministration of the individual components in healthy Chinese subjects in the fed state.
Incidence of adverse events | From Day 1 to Day 4, in Treatment period 1 and 2, respectively. An average of 11 to 18 days.
  To further assess the safety and tolerability of dapagliflozin/metformin XR FDC and coadministration of the individual components in healthy Chinese subjects in the fed state.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, MD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- Research Site, Suzhou, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Zhao X, Ning R, Hui A, Boulton DW, Tang W. Pharmacokinetic Variables of Dapagliflozin/Metformin Extended-release Fixed-dose Combination in Healthy Chinese Volunteers and Regional Comparison. Clin Ther. 2023 Aug;45(8):762-769. doi: 10.1016/j.clinthera.2023.06.012. Epub 2023 Jul 11. PMID 37442656